CLINICAL TRIAL: NCT06626308
Title: Early Biomarkers in Premanifest Huntington's Disease Gene Carriers: a Pilot Study
Acronym: BIO-MH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC24.0213; 2024-A01476-41 (Other: ID RCB)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Huntington Disease
Keywords: biomarkers; genetic carriers; brain functional MRI
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neuroimaging assessment (Experimental): visual stimulation protocol during functional MRI session
  Interventions: Other: brain functional MRI

INTERVENTIONS:
Other: brain functional MRI — visual protocol stimulation during brain functional MRI

SUMMARY:
The goal of this clinical trial is to investigate if new, early biomarkers of the disease are available in presymptomatic genetic carriers of Huntington's diesase compared to healthy subjects. The main questions it aims to answer are:

Does functional brain MRI is able to detect early biomarkers of the disease in genetic carriers? Does gait study by a virtual reality device can detect early biomarkers of the disease in genetic carriers? Researchers will compare genetic carriers and healthy subjects to see if new, early biomarkers of the disease can be detected .

DETAILED DESCRIPTION:
Huntington's disease (HD) is an autosomal dominant, neurodegenerative, fatal disease caused by a mutation in the hungtingtin (HTT) gene,1 manifesting with neurological, psychiatric and cognitive disorders. The disease causes a severe physical, functional and social impairment, with a great impact on patients' and their care-givers' quality of life. To date, the pathophysiology of HD remains largely unknown. Neuronal degeneration of basal ganglia plays a primary role in causing neuropsychiatric symptoms. Nevertheless, a cortical involvement has been evoked in the genesis of other symptoms of the disease, such as visual system disorders.2 To date only symptomatic treatment is available for motor and psychiatric issues in HD patients. The research field is now focused on investigation of genetic neuroprotective strategies to prevent the progression of the disease.3 The ideal therapeutic goal would be to start the treatment as soon as the disease becomes symptomatic, as the HD mutation is present since the birth. Unfortunately, the age and the symptoms at onset are very variable, mainly related to the mutation size4 but not only. Several other genetic and environmental factors are thought to play a role in the transition from the pre-symptomatic to the symptomatic stage, which remains largely unpredictable.5 Moreover, the diagnosis of symptomatic HD is traditionally based on motor symptoms onset (chorea, dystonia, bradykinesia, coordination issues).6 There are some evidence that subtle structural brain MRI alterations, mild cognitive and psychiatric issues may be present even in the pre-symptomatic stage, suggesting that the symptomatic phase could start before the onset of classical motor symptoms.7 Clinical studies using morphological and functional MRI have recently shown an early involvement of the visual cortex (area visual associative, lateral occipital cortex), which may explain the visuospatial function and visual perception disorders already observed at the pre-symptomatic and initial symptomatic stage of MH.8 The superior colliculus (SC) is a mesencephalic structure involved in the integration of visual stimuli, in the generation of oriented ocular saccades and attention tasks.9 An early dysfunction of SC has been shown in other diseases of the basal ganglia, such as Parkinson's disease (PD)10 and focal dystonia.11 This structure may also be early involved in the pathogenesis of visual disturbances and ocular saccadic changes described in HD.12 To date, there is no data regarding the functional state of SC in response to visual stimuli in HD.

Gait and balance issues in HD are common at the symptomatic stage of the disease, being a major risk of falls along with abnormal involuntary movements.13 They can be present at the early stage of the disease, with a mild severity. To date, no data are available about specific gait assessment in the pre-symptomatic HD carriers. Subtle gait issues resulting in spatiotemporal parameters alteration, not detectable with the standard clinical examination, could be present even in HD asymptomatic gene carriers. New technologies based on 3D virtual reality tools could be of great interest in the diagnosis of very early gait issues in pre-symptomatic HD subjects.

Cognitive issues are also common in HD, ranging from mild cognitive impairment in pre-manifest subjects14 to dementia in the advanced disease.15 Cognitive and emotional impairment is related to the basal ganglia degeneration in HD, progressively involving frontal and subcortical limbic regions.16 Eye-tracking data are known to be good markers of the orientation of attention. Recently, our team has shown that PD is associated in particular with dysfunction of the SC.10,17 At the same time, PD patients have difficulty producing and recognizing facial and vocal emotional expressions and are less reactive to negative stimuli than HS.18 As PD and HD share similar basal ganglia network dysfunctions, they could share also similar cognitive and emotional changes, which may be present from the onset of HD, due to structural and/or functional deficits in frontal and subcortical limbic areas. To date, no study has investigated emotional behavior and orientation reactions correlated with specific functional MRI (fMRI) protocol in pre-symptomatic HD carriers.

Objectives :

The primary objective of our study is to investigate the function of SC in response to visual stimulation using a fMRI in premanifest HD gene carriers (PMGC) compared to healthy subjects (HS). Our main hypothesis is the dysfunction of the SC at the pre-symptomatic stage of the disease (role of SC as an early biomarker of the disease).

Secondary objectives will be:

1. To study gait parameters using 3D virtual reality equipment in PMGC compared to HC, to demonstrate that they are abnormal at the pre-symptomatic stage of the disease.
2. To investigate the cognitive/emotional behavior in PMGC compared to HC, to demonstrate that it is abnormal at the pre-symptomatic stage of the disease.
3. To study the correlation between gait, neuroimaging, cognitive/emotional data and various clinical and neuropsychological variables.
4. To investigate potential pre-symptomatic subtypes profiles in HD carriers, based on neuroimaging, clinical, cognitive/emotional assessments correlation analysis.

Methodology :

Our study is a prospective, single-center, case-control, pilot study. Ten PMGC and ten age (+/- 5 years)- and sex-matched HS will be included. Main inclusion criteria will be: 1. For PMGC: HD diagnosis confirmed by genetic testing (CAG triplets ≥36 in HTT gene); Unified Huntington Disease Rating Scale19 Total Motor Score (UHDRS-TMS) ≤ 5; age 18-70 years old. 2. For HC: normal neurological examination; age 18-70 years old. Main exclusion criteria for both PMGC and HS will be: major ophthalmologic and psychiatric active diseases; cognitive impairment (Montreal Cognitive Assessment, MoCA score < 25/30); gait issues related to non-neurological conditions; contraindications to brain MRI.

Study design:

Selection of study population and inclusion in the study (V0). The PMGC will be selected in the Movement Disorders Unit of Grenoble University Hospital during a neuro-genetic consultation after genetic testing performed at the Service of Genetics at CHU Grenoble Alpes. HS will be recruited by means of advertisements published on the CNRS cognitive science website (http://www.risc.cnrs.fr/), and posted in the Service of Neurology, research laboratories belonging to UGA, and on the HD patients association website (https://huntington.fr). Informed consent to the study will be signed by the participants. Inclusion and exclusion criteria will be verified and the neurological assessment will be realized by an experienced neurologist in movement disorders.

Ophthalmologic visit (V1).The PMGC and the HS will perform an ophthalmological examination (measurement of visual acuity, fundus of the eye, visual field). The maximal time interval between V0 and V1 will be 1 month.

Neuropsychological assessment (V2). A complete neuropsychological assessment will be performed in PMGC by an experienced neuropsychologist in movement disorders, including: a. assessment of executive functions using frontal score, Stroop Delis-Kaplan, letter/number sequence (oral version of TMT); b. Memory assessment using WAIS IV, Corsi blocks, RL/R116 and Doors test; c. Assessment of instrumental functions with the BJLO-15 items, VOSP, BECS; d. Behavioural assessment with the BDI-II, LARS, SHAPS, STAI, UHDRS (psycho-behavioural part).

Functional MRI session (V3). Pre-symptomatic subjects and HS will perform an fMRI session. The time interval between V2 and V3 will be set between 2 weeks and 2 months. The fMRI acquisitions will be performed during 1 hour under visual stimulation, according to the protocol developed by our team.

Gait assessment (V4). The gait parameters of PGMC and HS will be assessed during 1 hour-visit using a special 3D equipment in the Movement Disorders Unit. The time interval between V3 and V4 will be set between 2 weeks and 2 months.

Cognitive/emotional assessment (V5). The study population will perform two different experimental sessions: one using eye-tracking for a task involving free exploration of emotional stimuli and the other using fMRI coupled with eye-tracking for tasks based on emotional feelings and the tendency to act. The time interval between V4 and V5 will be set between 2 weeks and 2 months.

After the V5, the study will end. Neuroimaging assessment The neuroimaging procedure includes: anatomical and perfusion brain MRI, and fMRI with a visual stimulation protocol.8 fMRI procedure. MRI acquisitions will be performed at the IRMaGE MRI facility in Grenoble using a whole-body 3-Tesla Philips Achieva MRI scanner equipped with a 32 channel SENSE head coil. Participants will be instructed to fixate a cross localized at the center of a screen in front of their eyes, on which the visual stimuli is presented to control ocular saccades. During each functional session, PRL and eye movements will be monitored using the ASL 6000 eye-tracker. To maintain and control the attention, each participant will be instructed to press a button when the orientation of the cross changes. The visual stimulation protocol comprises a series of achromatic checkerboards with four levels of luminance contrast (1%, 3%, 5%, and 9%) and flashing at a frequency of 4Hz on a grey background. Each fMRI run is composed of four 12-s blocks of visual stimulation, one for each contrast (Figure 1), and five 12-s fixation intervals. The complete functional MRI session is composed of nine scanning runs, leading to 36 randomized block-presentations of each luminance contrast level. The cardiac signal is indirectly recorded based on the hemodynamic pulse at fingertip using the pulse plethysmography unit attached to the MRI scanner.

MRI sequences. Functional, anatomical, and perfusion measurements will be performed during each MRI session. For functional scans, a standard gradient echo planar imaging sequence will be used. Twenty-five slices (1.5 mm) will be acquired covering the SC, the lateral geniculate nucleus (LGN) and the primary visual area cortex (V1). High-resolution structural images will be acquired using T1-weighted 3D MP-RAGE and FGATIR sequences and used for manual delineation of our regions-of-interest (ROI) (Figure 2). A whole-brain pseudo-continuous arterial spin labeling (ASL) sequence will be used to measure brain tissue perfusion.

Gait assessment

The gait protocol assessment will be performed using a 3D specific equipment developed by Social Dreams® enterprise. This equipment is already available on the market, with CE authorization (www.socialdreams.fr). It has been applied in ongoing clinical studies investigating gait function and cognitive stimulation in patients with Alzheimer's disease in the Geriatric Service of the CHU of Lyon, France. Data not yet published). The equipment includes:

1. PERCEPTION NEURON3 (PN3, figure 3): a body multisensor-motion capture-integrated suite, able to capture any body movement, with no constraints on space, lighting or environment. The PN3 " Body Kit " includes: PN3 Body Sensors (17); PN3 Spare Sensor (1); PN3 USB Transceiver (1); Body Straps (1 set); Charging Docks (3); Axis Studio License dongle (1); USB-A to USB-C cable (3); USB-A Male to USB-C Female; Axis Neuron capture and recording software.
2. PICOG3 (figure 4): a 3DOF VR headset with 4K screen and integrated audio system, with six degrees of freedom, able to track the movements of both head and body, and to reproduce them in Virtual Reality with realistic accuracy, with no external sensors required. The kit includes also: a TP-LINK TL-WR902AC Routeur sans fil Dual-Band Wi-Fi AC (AC430+ N300); a tactile Tablette Lenovo Tab P11 - 11'' 2K LCD (Processeur Qualcomm Snapdragon 662 8Coeurs, 4 Go de RAM, UFS 64 Go, Qualcomm Adreno 610 GPU, Android 10, 4G LTE, WiFi+Bluetooth); two joysticks.

Gait spatiotemporal parameters will be assessed during three different session (5 minutes/session). A pause of 5 minutes between each session will be performed. Three different 3D scenarios will be created, with increasing gait difficulty levels (obstacles, turns…), and projected using the PICOG3 headset for each of the three sessions.

Cognitive/emotional assessment

1. The fMRI session will be performed at the IRMaGE MRI facility in Grenoble (see neuroimaging assessment).

   Stimuli: The fMRI task will involve the individual visualisation of colour photographs of natural scenes. These photographs will be taken from the image database selected for the eye-tracking study described below. They will include 60 negative stimuli, 60 positive stimuli and 60 neutral stimuli divided into 2 groups of stimuli: one group (gr1High) will include high-activation negative and positive emotional stimuli and neutral stimuli and the other group (gr2Blow) will include low-activation negative and positive emotional stimuli and neutral stimuli.

   The stimuli will be projected onto a screen at the back of the magnet, which participants will be able to view via a mirror attached to the head's radio-frequency antenna.

   Experimentation. The experiment will last a maximum of 1 hour, including set-up time, sessions and breaks. Each participant will perform 2x2 functional MRI scans (total duration 22 minutes): 2 scans will be performed with high-activation stimuli (grp1High) and 2 others with low-activation stimuli (grp2Blow). The order of the scans of the 2 types of stimuli (high and low activation) will be alternated between PMGC and HS. Each scan will present a succession of photographs of natural scenes of negative, positive and neutral valence (30 of each) and null events (fixation cross replacing the photograph in the trial) according to a mixed paradigm. Each photograph will be presented for 1 second, interspersed with a cross of fixation lasting 1500 ms. The 2 scans of each type of stimulus will be distinguished by the nature of the task to be performed: emotional task or action tendency task. In the emotional task, the participant will have to indicate his emotional experience for each scene as quickly and accurately as possible as soon as the photograph appears, i.e. he will have to decide, for each trial, whether the scene is unpleasant, pleasant or neutral (no emotion) by pressing the corresponding response button. During the action tendency task, the participant will have to indicate the action he would take if he were involved in this situation in reality as quickly and accurately as possible as soon as the photograph appears, i.e. he will have to decide, for each trial, whether he would move away (avoid), approach, or not move, by pressing the corresponding response button. Each task will involve 3 response choices corresponding to 3 button choices. The assignment of the buttons to the 3 emotions (emotional task) or to the 3 action tendencies (action task) will be indicated to the participants beforehand and will be counterbalanced between the participants. The participant's responses and response times will be recorded for each trial. Participants will be familiarized with each task beforehand, using different training trials to those used in the experiment. The brain regions of interest selective to emotional processing will be functionally identified for each participant by performing a 5-minute 'localizer' scan. Participants will view photographs and scrambles (random assembly of scene pieces) of natural scenes of negative valence (scenes of mutilation) and neutral valence (environments, houses) in separate blocks of a block paradigm and will be asked to indicate when 2 identical photographs follow each other. Throughout the fMRI acquisitions (except during the localizer), eye positions and movements will be recorded using an oculometer. The calibration procedure before each functional scan and during the experiment will be identical to that described in the previous eye-tracking experiment. Between the 2 series of scans, a 4-minute high-resolution anatomical MRI will be acquired in order to normalise the MRI data (registration) between the scans of the same participant and between the participants. The experimental run in the MRI will be completed by the acquisition of an 8-minute perfusion image and an 8-minute diffusion imaging (DTI) optimized for the visual system. The perfusion image will allow us to ensure that the BOLD signal is interpreted under good perfusion conditions. During the anatomical MRI and the DTI, participants will watch a film to pass the time or may close their eyes if they wish. At the end of the MRI acquisitions, after a break, the participant will perform a final subjective evaluation task of emotional photographs (200), including those used in the fMRI study, over a maximum of 20 minutes. The task will involve accurately assessing the level of valence, activation and action tendency of each photograph. This assessment will help refine the analyses of the fMRI data and establish a normative image database for de novo Parkinson's patients for future studies.
2. Eyetracker assessment: Eye movements will be measured during MRI sessions using the MRI-compatible EyeLink 1000 plus (SR Research). Pupillary diameter, saccades and blinks will be quantified using EyeLink software. The same equipment is available outside MRI for behavioral control measurements.

Statistical analysis The primary outcome of the study is the measurement of BOLD (Blood Oxygen Level Dependent) signal changes using fMRI (3 Tesla), in two subcortical regions, SC, LGN, and V1 in response to visual stimuli, in PMGC compared to HS. Analysis of the BOLD signal for these three ROIs will be done for both hemispheres together. A Bonferroni correction between the luminance levels will be performed. The Friedman test will be used to analyse the effects of luminance contrast changes of each ROI within each group. The Mann-Whitney test will be used to compare between groups the response of each ROI for each luminance contrast. Analysis of variance (ANOVA) will be used to assess the cerebral perfusion data within and between groups and regions of interests (SC, LGN and V1). Because the SC is also involved in the control of voluntary and reflexive ocular saccades, we will investigate eye movements during the MRI study. The number of saccades for each participant will be computed from oculomotor signal analysis. The number of successful detections of the central cross changes during the attentional task between the two groups will be analysed using the Mann-Whitney test.

With respect to the sample size, our previous study demonstrated that, when using our specific fMRI paradigm on 20 individuals, the effect size was sufficient to allow a robust statistical analysis of the BOLD signal modulation in the visual structures of interest8. A power analysis performed in the two study groups shows that the number of subjects involved could allow drawing valid conclusions (G power = 0.94). All statistical analysis will be performed by the Neuroimaging Team (IRMAGE research platform, GIN).

The secondary outcomes are:

1. Measurement of gait spatiotemporal parameters (stance time, swing time, double support time, stride time, stride length, and step length) during the three different gait challenging 3D visual scenarios in PMGC compared to HS. Analysis of these data will be performed using dedicated softwares Axis Neuron and a musculoskeletal analysis software package developed in MATLAB®.
2. Comparison of behavioural measures, reaction times and congruent response rates between PMGC and HS.

   Eye-tracking session: Mean first saccade orientation rate and mean first saccade latency will be statistically analysed for each emotional valence according to activation level and pair type using a repeated measures ANOVA with population (patients and healthy controls) as a between-subjects variable and activation level (HIGH and LOW) and stimulus valence according to pairs (NEG with positive, NEG with neutral, POS with negative, POS with neutral, NEU with positive and NEU with negative) as within-subjects variables. Comparisons of means were evaluated using a Tukey post-hoc test. For all statistical analyses, the significance threshold will be 0.05. As for the other oculomotor parameters, two levels of analysis will be considered: analysis over the total duration of presentation of the pairs of stimuli and by time period. For each participant and each experimental condition (types of pairs, intensity of stimuli), the mean values of the different parameters considered (duration of fixations, rate and dispersion of eye saccades for each stimulus of each pair) will be calculated over the total duration of presentation of the pairs of scenes and analysed statistically for each emotional valence (negative, positive and neutral) according to pair type and stimulus activation level using a repeated measures ANOVA with population (patients and healthy controls) as the between-subjects variable and activation level (HIGH and LOW) and stimulus valence according to pairs (NEG with positive, NEG with neutral, POS with negative, POS with neutral, NEU with positive and NEU with negative) as the within-subjects variables. Comparisons of means were evaluated using a Tukey post-hoc test. For all statistical analyses, the significance threshold will be 0.05.

   Eye-tracking measurements from the fMRI study: parameters similar to eye-tracking study 1 will be extracted, such as the latency of the first saccade and the rate and duration of fixations for each stimulus. They will be analysed statistically using a repeated measures ANOVA with the population (patients vs controls) as the between-subjects variable and the task (emotional and action tendency), the activation level (high and low) and the valence of the stimuli (negative, positive, neutral) as the within-subjects variables. Comparisons of means were evaluated using a Tukey post-hoc test. For all statistical analyses, the significance threshold will be 0.05. Correlation analyses will also be considered between eye-tracking data and fMRI data. The eye-tracking data will also allow us to eliminate neural correlates of activation linked to palpebral blinks.

   Behavioural data: Reaction times (in ms) and the percentage of "correct" responses will be analysed statistically (ANOVAs, Tuckey post-hoc tests) with the group of participants (patients, controls) as a within-subjects factor and the task, valence and activation level of the stimuli as between-subjects factors.
3. Data Correlation study The data from the various assessments (gait, neuroimaging, cognitive/emotional) will be evaluated in relation to the various clinical variables (e.g. age, motor scores, etc.) and neuropsychological variables using correlation analyses. The correlative study of neuropsychological scores with structural and physiological biomarkers may help to identify new ways of discriminating the individual profiles of pre-symptomatic HD subjects.
4. Estimation of subtypes of pre-symptomatic HD subjects:

Other analyses based on statistical classification methods will be considered on the basis of the various data acquired (functional, structural, effective connectivity, oculomotor activity data, etc.) in order to identify characteristics or indexes of characteristics that discriminate subtypes of pre-symptomatic HD subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. For PMGC: HD diagnosis confirmed by genetic testing (CAG triplets ≥36 in HTT gene); Unified Huntington Disease Rating Scale19 Total Motor Score (UHDRS-TMS) ≤ 5; age 18-70 years old. 2. For HC: normal neurological examination; age 18-70 years old.

Exclusion Criteria:

* Main exclusion criteria for both PMGC and HS will be: major ophthalmologic and psychiatric active diseases; cognitive impairment (Montreal Cognitive Assessment, MoCA score < 25/30); gait issues related to non-neurological conditions; contraindications to brain MRI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brain functional MRI biomarker investigation | from the enrollement to the end of the investigation: 2 months
  Measurement of BOLD (Blood Oxygen Level Dependent) signal changes using fMRI (3 Tesla), in two subcortical regions, SC, LGN, and V1 in response to visual stimuli, in PMGC compared to HS.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France